CLINICAL TRIAL: NCT05639907
Title: A Comparison of Miniscrew Stability and Peri-implant Inflammation When Precoated With Antimicrobial Quaternary Ammonium Compound K21 vs Ethanol Control in Orthodontic Patients: a Triple-blind, Split-mouth, Randomized Controlled Clinical Trial
Brief Title: Miniscrew Stability and Peri-implant Inflammation When Precoated K21 vs Ethanol Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 22-1579
Record Dates: First submitted 2022-11-15; First posted 2022-12-07 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Inflammation Caused by the Placement of a Temporary Anchorage Device
Keywords: TAD; inflammation; orthodontics
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: Split mouth
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: There will be random allocation established, such that as a study participant is enrolled the clinician will receive a numbered envelope that contains the information for which TAD placement site will receive a TAD coated with solution A or B. The identification of Solution A or B is kept secret in an envelope stored in the office of the Chair of the Orthodontic Department (U Colo, Sch Dent Med). The patient, clinical operator, Investigator and Outcomes assessor is not aware which solution (A or B) is the experimental or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- K21 Cavity cleanser-coated TAD (Experimental): A TAD to be placed is coated with K21 solution. The solution is allowed to evaporate to dryness, leaving a K21-rich film. The TAD is placed following the University TAD placement protocol.
  Interventions: Device: K21 Cavity cleanser
- Ethanol Control (Placebo Comparator): A TAD to be placed is coated with ethanol solution. The solution is allowed to evaporate to dryness (no residue is expected). The TAD is placed following the University TAD placement protocol.
  Interventions: Device: Ethanol control

INTERVENTIONS:
Device: K21 Cavity cleanser — K21 Cavity cleanser is rinsed over the TAD and allowed to dry. The TAD is placed where needed for orthodontic therapy following the Department of Orthodontics protocols.
  Arms: K21 Cavity cleanser-coated TAD
Device: Ethanol control — Ethanol is rinsed over the TAD and allowed to dry. The TAD is placed where needed for orthodontic therapy following the Department of Orthodontics protocols.
  Arms: Ethanol Control

SUMMARY:
To determine if coating miniscrews with K21 would increase the success rate of orthodontic miniscrews by reducing adjacent tissue inflammation.

DETAILED DESCRIPTION:
The study design is a split mouth study where 2 miniscrews, one pretreated with K21 the other pretreated (experimental) with ethanol (placebo) are placed in the mouth for orthodontic therapy. All participants will receive 2 or more orthodontic miniscrews with equal numbers of experimental and control pretreatment solutions. Mobility will be assessed at the 4 and 8 week follow up appointments by gentle manipulation with cotton pliers. Clinical success will be defined as maintenance of stability for a period of 8 weeks. Peri-implant inflammation will be assessed at follow up appointments by looking for signs of soft-tissue inflammation (redness, swelling) where possible.

ELIGIBILITY:
Inclusion Criteria:

1. Good general health, with no significant medical findings
2. Requiring at least two miniscrews in their treatment plans (i.e., most participants will have two miniscrews, but some may receive four or six as indicated by their individual treatment plan)
3. Miniscrew pairs indicated with comparable anatomical positions and comparable mechanics (direct vs. indirect anchorage).

Exclusion Criteria:

1. Recent or ongoing use of antiresorptive pharmacological agents contraindicating the use of orthodontic miniscrews
2. Less than 12 years of age
3. Heavy tobacco use (>10 cigarettes/day)
4. Peri-implant tissues must be observable at follow-up appointments
5. Being unable or unwilling to consent to the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
TAD motility | 8 weeks
  The motility of a TAD is evaluated by gentle manipulation with cotton pliers. Clinical failures will be defined as a mobility greater than or equal to 1mm. Clinical success will be defined as maintenance of stability for a period of 8 weeks.
Peri-implant inflammation | 8 weeks
  Inspection for signs of soft-tissue inflammation (redness, swelling) immediately around the TAD. The Loe-Silness Index scale will be used to assess any inflammation. The Loe-Silness Index scale is between 0 and 3 where a 0 is normal soft tissue, 1 is mild inflammation where the tissue color is slightly red and the tissue does not bleed upon probing, 2 is moderate inflammation where the tissue color is red with edema and bleeds upon probing, and 3 is severe inflammation where the tissue bleeds with little or no probing has edema and has ulcers.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado School of Dental Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alharbi F, Almuzian M, Bearn D. Miniscrews failure rate in orthodontics: systematic review and meta-analysis. Eur J Orthod. 2018 Sep 28;40(5):519-530. doi: 10.1093/ejo/cjx093. PMID 29315365
- [Result] Cheng SJ, Tseng IY, Lee JJ, Kok SH. A prospective study of the risk factors associated with failure of mini-implants used for orthodontic anchorage. Int J Oral Maxillofac Implants. 2004 Jan-Feb;19(1):100-6. PMID 14982362
- [Result] Daood U, Matinlinna JP, Pichika MR, Mak KK, Nagendrababu V, Fawzy AS. A quaternary ammonium silane antimicrobial triggers bacterial membrane and biofilm destruction. Sci Rep. 2020 Jul 3;10(1):10970. doi: 10.1038/s41598-020-67616-z. PMID 32620785
- [Result] Kok ESK, Lim XJ, Chew SX, Ong SF, See LY, Lim SH, Wong LA, Davamani F, Nagendrababu V, Fawzy A, Daood U. Quaternary ammonium silane (k21) based intracanal medicament triggers biofilm destruction. BMC Oral Health. 2021 Mar 12;21(1):116. doi: 10.1186/s12903-021-01470-x. PMID 33711992
- [Result] Meghil MM, Rueggeberg F, El-Awady A, Miles B, Tay F, Pashley D, Cutler CW. Novel Coating of Surgical Suture Confers Antimicrobial Activity Against Porphyromonas gingivalis and Enterococcus faecalis. J Periodontol. 2015 Jun;86(6):788-94. doi: 10.1902/jop.2015.140528. Epub 2015 Feb 23. PMID 25703732